CLINICAL TRIAL: NCT01551758
Title: A 12-month, Open Label, Randomised, Effectiveness Study to Evaluate Fluticasone Furoate (FF, GW685698)/Vilanterol (VI, GW642444) Inhalation Powder Delivered Once Daily Via a Novel Dry Powder Inhaler (NDPI) Compared With the Existing COPD Maintenance Therapy Alone in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Randomised Effectiveness Study Comparing Fluticasone Furoate (FF, GW685698)/Vilanterol (VI, GW642444) With Standard Treatment in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115151
Record Dates: First submitted 2012-03-01; First posted 2012-03-13 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Exacerbation; Adult; COPD; Respiratory
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FF/VI (Experimental): once daily via a Novel Dry Powder Inhaler
  Interventions: Drug: FF/VI
- Existing Maintenance Therapy (Other): Existing Maintenance Therapy:
  * Long acting bronchodilator therapy alone
  * ICS alone or in combination with a long acting bronchodilator
  * Triple maintenance therapy
  Interventions: Other: Existing Maintenance Therapy

INTERVENTIONS:
Drug: FF/VI — FF/VI
  Arms: FF/VI
Other: Existing Maintenance Therapy — Existing Maintenance Therapy:
  * Long acting bronchodilator therapy alone
  * ICS alone or in combination with a long acting bronchodilator
  * Triple maintenance therapy
  Arms: Existing Maintenance Therapy

SUMMARY:
This study is designed to compare the effectiveness and safety of Fluticasone Furoate/Vilanterol Inhalation Powder (100mcg Fluticasone Furoate ((FF), GW685698)/25mcg Vilanterol ((VI), GW642444)) delivered once daily via a Novel Dry Powder Inhaler (NDPI) compared with the existing COPD maintenance therapy over twelve months in subjects diagnosed with COPD. This is a Phase III multi-centre, randomised open label study. Subjects who meet the eligibility criteria are randomised and will enter a 12 month treatment period.

DETAILED DESCRIPTION:
This is a Phase III multi-centre, randomised open label study performed in subjects followed in primary care who have a diagnosis of and receive regular treatment for COPD in a localised geographical region of the UK

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

1. Type of subject: Subjects with documented GP diagnosis of COPD, and currently receiving maintenance therapy
2. Informed consent: Subjects must be able to provide informed consent, have their consent signed and dated. Subjects must be able to complete the electronic subject questionnaires or allow a proxy to do so on their behalf.
3. Gender and Age: Male or female subjects aged ≥40 years of age at Visit 1 A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms. However in questionable cases, a blood sample with FSH > 40MIU/ml and estradiol <40pg/ml (<140 pmol/L) is confirmatory. Or child bearing potential has a negative urine pregnancy test at Visit 2, and agrees to one of the highly effective and acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label and the instructions of the physician for the duration of the study - Visit 2 to the end of the study).
4. Subjects with Exacerbation History
5. Current COPD Maintenance Therapy

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

1. Subjects with any life threatening condition (e.g. low probability (in the opinion of the GP/Investigator) of 12 month survival due to severity of COPD or co-morbid condition) at the point of entry into the study.
2. Other diseases/abnormalities: Subjects with historical or current evidence of uncontrolled or clinically significant disease. Significant is defined as any disease that, in the opinion of the GP/ Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
3. Subjects with unstable COPD, defined as the occurrence of the following in the 2 weeks prior to Visit 2:

   - Acute worsening of COPD that is managed by the subject with corticosteroids or antibiotics or that requires treatment prescribed by a physician.
4. Chronic user of oral corticosteroids: Subjects who, in the opinion of the GP/Investigator, are considered to be a chronic user of oral corticosteroids for respiratory or other indications (if unsure discuss with the medical monitor prior to screening)
5. Drug/food allergy: Subjects with a history of hypersensitivity to any of the study medications (e.g., beta-agonists, corticosteroid) or components of the inhalation powder (e.g., lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the GP/ Investigator, contraindicates the subject's participation will also be excluded.
6. Investigational Medications: A subject must not have used any investigational drug treatment within 30 days prior to Visit 2 or within five half-lives (t½) of the prior investigational study (whichever is the longer of the two).
7. Subjects who plan to move away from the geographical area where the study is being conducted during the study period and/or if subjects have not consented to their medical records being part of the electronic medical records database that is operational in the Salford area.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2802 (Actual)
Dates: Start 2012-03-13 (Actual); Primary Completion 2015-11-24 (Actual); Study Completion 2015-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (44):
- United Kingdom (44):
  - GSK Investigational Site, Altrincham, Cheshire
  - GSK Investigational Site, Bowdon, Cheshire
  - GSK Investigational Site, Cheadle, Cheshire
  - GSK Investigational Site, Cheadle Hulme, Cheshire
  - GSK Investigational Site, Edgeley, Cheshire
  - GSK Investigational Site, Gatley, Cheshire
  - GSK Investigational Site, Heald Green, Cheshire
  - GSK Investigational Site, Sale, Cheshire
  - GSK Investigational Site, Stockport, Cheshire
  - GSK Investigational Site, Timperley, Cheshire
  - GSK Investigational Site, Altrincham, Greater Manchester
  - GSK Investigational Site, Broadway, Davyhulme, Greater Manchester
  - GSK Investigational Site, Irlam, Greater Manchester
  - GSK Investigational Site, Irlam, Manchester, Greater Manchester
  - GSK Investigational Site, Manchester, Greater Manchester
  - GSK Investigational Site, Newall Green, Greater Manchester
  - GSK Investigational Site, Northenden, Greater Manchester
  - GSK Investigational Site, Northern Moor, Greater Manchester
  - GSK Investigational Site, Pendlebury, Greater Manchester
  - GSK Investigational Site, Pendlebury, Manchester, Greater Manchester
  - GSK Investigational Site, Salford, Greater Manchester
  - GSK Investigational Site, Salford, Manchester, Greater Manchester
  - GSK Investigational Site, Stretford, Greater Manchester
  - GSK Investigational Site, Timperley, Greater Manchester
  - GSK Investigational Site, Withington, Greater Manchester
  - GSK Investigational Site, Wythenshawe, Greater Manchester
  - GSK Investigational Site, Cadishead, Manchester
  - GSK Investigational Site, Cheadle
  - GSK Investigational Site, Eccles
  - GSK Investigational Site, Eccles, Manchester
  - GSK Investigational Site, Ellenbrook, Manchester
  - GSK Investigational Site, Irlam, Manchester
  - GSK Investigational Site, Irlam, Salford
  - GSK Investigational Site, Little Hulton, Manchester
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Pendlebury, Manchester
  - GSK Investigational Site, Salford
  - GSK Investigational Site, Salford, Manchester
  - GSK Investigational Site, Stockport
  - GSK Investigational Site, Swinton
  - GSK Investigational Site, Swinton, Manchester
  - GSK Investigational Site, Walkden, Manchester
  - GSK Investigational Site, Worsley, Manchester
  - GSK Investigational Site, Wythenshawe

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Vestbo J, Waterer G, Leather D, Crim C, Diar Bakerly N, Frith L, Jacques L, Harvey C, Satia I, Woodcock A; Salford Lung Study Investigators. Mortality after admission with pneumonia is higher than after admission with an exacerbation of COPD. Eur Respir J. 2022 May 19;59(5):2102899. doi: 10.1183/13993003.02899-2021. Print 2022 May. PMID 35273031
- [Derived] Bakerly ND, Browning D, Boucot I, Crawford J, McCorkindale S, Stein N, New JP. The impact of fluticasone furoate/vilanterol on healthcare resource utilisation in the Salford Lung Study in chronic obstructive pulmonary disease. Ther Adv Respir Dis. 2021 Jan-Dec;15:17534666211001013. doi: 10.1177/17534666211001013. PMID 33781142
- [Derived] Sperrin M, Webb DJ, Patel P, Davis KJ, Collier S, Pate A, Leather DA, Pimenta JM. Chronic obstructive pulmonary disease exacerbation episodes derived from electronic health record data validated using clinical trial data. Pharmacoepidemiol Drug Saf. 2019 Oct;28(10):1369-1376. doi: 10.1002/pds.4883. Epub 2019 Aug 5. PMID 31385428
- [Derived] Bakerly ND, Woodcock A, Collier S, Leather DA, New JP, Crawford J, Harvey C, Vestbo J, Boucot I. Benefit and safety of fluticasone furoate/vilanterol in the Salford Lung Study in chronic obstructive pulmonary disease (SLS COPD) according to baseline patient characteristics and treatment subgroups. Respir Med. 2019 Feb;147:58-65. doi: 10.1016/j.rmed.2018.12.016. Epub 2019 Jan 10. PMID 30704700
- [Derived] Woodcock A, Boucot I, Leather DA, Crawford J, Collier S, Bakerly ND, Hilton E, Vestbo J. Effectiveness versus efficacy trials in COPD: how study design influences outcomes and applicability. Eur Respir J. 2018 Feb 21;51(2):1701531. doi: 10.1183/13993003.01531-2017. Print 2018 Feb. PMID 29467200
- [Derived] Vestbo J, Leather D, Diar Bakerly N, New J, Gibson JM, McCorkindale S, Collier S, Crawford J, Frith L, Harvey C, Svedsater H, Woodcock A; Salford Lung Study Investigators. Effectiveness of Fluticasone Furoate-Vilanterol for COPD in Clinical Practice. N Engl J Med. 2016 Sep 29;375(13):1253-60. doi: 10.1056/NEJMoa1608033. Epub 2016 Sep 4. PMID 27593504
- [Derived] Bakerly ND, Woodcock A, New JP, Gibson JM, Wu W, Leather D, Vestbo J. The Salford Lung Study protocol: a pragmatic, randomised phase III real-world effectiveness trial in chronic obstructive pulmonary disease. Respir Res. 2015 Sep 4;16(1):101. doi: 10.1186/s12931-015-0267-6. PMID 26337978
- [Derived] New JP, Bakerly ND, Leather D, Woodcock A. Obtaining real-world evidence: the Salford Lung Study. Thorax. 2014 Dec;69(12):1152-4. doi: 10.1136/thoraxjnl-2014-205259. Epub 2014 Mar 6. PMID 24603195
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 115151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicentre, randomized, stratified, open-label study to evaluate the effectiveness and safety of fluticasone fuorate (FF)/vilanterol (VI) in participants followed in primary care who had a diagnosis of and received regular treatment for Chronic Obstructive Pulmonary Disease (COPD).
Pre-assignment Details: Participants (par.) were randomized 1:1 to receive 1 inhalation of FF/VI 100 microgram (mcg)/25 mcg once daily (QD) or continued their existing maintenance therapy for 12 months. 2802 par. were randomized (3 par. randomized to the FF/VI arm did not receive study medication). A total of 2799 par. comprised the Intent to Treat (ITT) Population.
Groups:
- Usual Care: Participants continued their existing maintenance therapy that included one of the following: an inhaled corticosteroid (ICS) alone or Long Acting Beta Agonist (LABA) alone or Long Acting Muscarinic Antagonist (LAMA) alone or combination of any two (ICS+LABA/ ICS+LAMA/ LABA+LAMA) or triple therapy (ICS+LABA+LAMA) at the appropriate dosing schedule, for 12 months
- Fluticasone Furoate (FF)/Vilanterol (VI) 100 mcg/25 mcg: Participants were prescribed one inhalation of fluticasone furoate /vilanterol (FF/VI) 100 mcg/25 mcg via dry powder inhaler (DPI) once daily in the morning for 12 months in lieu of existing maintenance therapy. Participants on previous triple therapy received LAMA therapy additionally.
Period: Overall Study
Arm/Group | Usual Care | Fluticasone Furoate (FF)/Vilanterol (VI) 100 mcg/25 mcg
Started | 1403 | 1396
Completed | 1309 | 1291
Not Completed | 94 | 105
Not completed — Adverse Event | 29 | 43
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 5 | 6
Not completed — Met Protocol-defined stopping criteria | 8 | 10
Not completed — Lost to Follow-up | 29 | 25
Not completed — Physician Decision | 9 | 3
Not completed — Withdrawal by Subject | 14 | 17

BASELINE CHARACTERISTICS:
Groups:
- FF/VI 100 mcg/25 mcg: Participants were prescribed one inhalation of fluticasone furoate/vilanterol (FF/VI) 100 mcg/25 mcg via dry powder inhaler (DPI) once daily in the morning for 12 months in lieu of existing maintenance therapy. Participants on previous triple therapy received LAMA therapy additionally.
- Total: Total of all reporting groups
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg | Total
Number analyzed (Participants) | 1403 | 1396 | 2799
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (9.93) | 66.6 (9.90) | 66.7 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 671 | 698 | 1369
  Male | 732 | 698 | 1430
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3 | 5 | 8
  Asian-Central/South Asian Heritage | 5 | 6 | 11
  Asian-East Asian Heritage | 1 | 0 | 1
  Asian-South East Asian Heritage | 1 | 0 | 1
  White-Arabic/North African Heritage | 1 | 3 | 4
  White-White/Caucasian/European Heritage | 1387 | 1376 | 2763
  Mixed Race | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Annual Rate of Moderate or Severe COPD Exacerbations
Description: Mean annual rate of moderate or severe COPD exacerbations during treatment were assessed. Moderate exacerbation: participant received exacerbation-related prescription of oral corticosteroids and/ or antibiotic (with/without National Health Service [NHS] contact) not requiring hospitalisation. Severe exacerbation: an exacerbation-related hospitalisation. Analysis method was Generalised Linear Model (GLM) assuming the negative binomial distribution with a log-link function and logarithm of time on treatment as an offset variable, adjusted for randomized treatment, baseline COPD maintenance therapy per randomisation stratification, number of moderate/severe COPD exacerbations in previous year and smoking status at baseline. Intent to treat (ITT) population: all randomised participants who received a prescription of study medication. Primary Efficacy Analysis Population: all ITT participants who had at least one moderate/severe exacerbation in the year prior to randomization
Time Frame: Up to 54 weeks
Population: Primary Efficacy Analysis Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Groups:
- FF/VI 100 mcg/25 mcg: Existing Maintenance Therapy:
  * Long acting bronchodilator therapy alone
  * ICS alone or in combination with a long acting bronchodilator
  * Triple maintenance therapy
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1134 | 1135
Exacerbations per participant per year | 1.90 [1.80 to 2.01] | 1.74 [1.65 to 1.84]
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p = 0.025, Generalized Linear Model; Adjusted treatment ratio = 0.92, 95% CI 2-sided [0.85 to 0.99]

2. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) of Pneumonia During the Study
Description: Incidence of SAE of pneumonia was defined for each randomized treatment group as the proportion (number) of participants in that group who experienced at least one SAE of pneumonia in the Pneumonia Adverse Event of Special Interest subgroup during the treatment period (from start date of exposure to stop date of exposure + 28 days). Non-inferiority is demonstrated if the upper limit of the two-sided 95% confidence interval for the incidence ratio is less than 2. Serious Adverse Events of pneumonia are defined by the Pneumonia Special Interest Group, which for SAEs of pneumonia collected for these subjects includes the following preferred terms: Pneumonia, Pneumonia aspiration, Aspergillus infection, Empyema, Pneumonia streptococcal, Pneumonitis, Pulmonary tuberculosis.
Time Frame: Up to 58 weeks
Population: The Intent-to-Treat (ITT) Population: Defined as all participants who were randomised and received at least one prescription of study medication
Measure: Number; unit: Participants
Groups:
- FF/VI 100 mcg/25 mcg: Participants were prescribed one inhalation of fluticasone furoate /vilanterol (FF/VI) 100 mcg/25 mcg via dry powder inhaler (DPI) once daily in the morning for 12 months in lieu of existing maintenance therapy. Participants on previous triple therapy received LAMA therapy additionally.
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 83 | 94
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Non-Inferiority or Equivalence — Non-inferiority is demonstrated if the upper limit of the two-sided 95% confidence interval for the incidence ratio is less than 2; Incidence ratio = 1.1, 95% CI 2-sided [0.9 to 1.5] — Calculated as % of participants who had at least one SAE of pneumonia in the FF/VI group divided by the % of participants who had at least one SAE of pneumonia in the Usual Care group

3. Secondary Outcome: Mean Number of Serious Adverse Events of Pneumonia During the Study
Description: The mean number of SAE of pneumonia over the treatment period (from first date of exposure to last date of exposure + 28 days was calculated. Analysis was performed using a negative binomial regression model with covariates of randomised treatment and with logarithm of time on treatment as an offset variable.
Time Frame: Up to 58 weeks
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Mean Number of SAE
Groups:
- FF/VI 100 mcg/25 mcg: Participants were prescribed one inhalation of fluticasone fuorate /vilaneterol (FF/VI) 100 mcg/25 mcg via dry powder inhaler (DPI) once daily in the morning for 12 months in lieu of existing maintenance therapy. Participants on previous triple therapy received LAMA therapy additionally.
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Mean Number of SAE | 0.07 [0.06 to 0.09] | 0.08 [0.06 to 0.09]
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority or Other; p = 0.632, Generalized linear model; Adjusted treatment ratio = 1.08, 95% CI 2-sided [0.79 to 1.47]

4. Secondary Outcome: Time to the First Serious Adverse Event of Pneumonia Occuring in a Year
Description: The analysis method was a Cox proportional hazards model adjusted for randomized treatment. Analyses included those on-treatment SAEs of pneumonia that had an onset over the first 364 days of exposure, as defined. Participants who did not have an SAE of pneumonia during the first 364 days of the treatment period (start date of exposure to end date of exposure + 28 days were considered censored. Number of participants with event is presented.
Time Frame: Up to 52 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 80 | 89
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p = 0.439, Cox proportional hazards model; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.83 to 1.52]

5. Secondary Outcome: Number of COPD-related Secondary Care Contacts Expressed as Least Square Mean
Description: A COPD-related secondary care contact was defined as an inpatient admission or a specialist outpatient visit or an accident & emergency (A&E) contact. A participant with an A&E contact and subsequent inpatient admission was considered to have had two healthcare contacts. Inpatient admissions recorded at two hospitals on the same day, this was counted as a single (inpatient admission) secondary care contact. COPD-related contacts were identified using predefined lists of ICD-10 codes, specialty descriptions and diagnosis codes recorded in the patients electronic health record (EHR). GLM assuming the negative binomial distribution with log-link function and logarithm of time on treatment as an offset variable and adjusted for randomised treatment, baseline COPD maintenance therapy per randomisation stratification, number of moderate/severe COPD exacerbations in the previous year to randomisation and smoking status at baseline.
Time Frame: Up to 54 weeks
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Contacts per participant per year
Groups:
- FF/VI 100 mcg/25 mcg: ExParticipants were prescribed one inhalation of fluticasone fuorate /vilaneterol (FF/VI) 100 mcg/25 mcg via dry powder inhaler (DPI) once daily in the morning for 12 months in lieu of existing maintenance therapy. Participants on previous triple therapy received LAMA therapy additionally.
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Contacts per participant per year | 1.48 [1.30 to 1.67] | 1.57 [1.39 to 1.78]
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p = 0.488, Generalized linear model; Adjusted treatment ratio = 1.06, 95% CI 2-sided [0.89 to 1.27]

6. Secondary Outcome: Number of COPD-related Primary Care Contacts Expressed Using Least Square Mean
Description: A COPD-related primary care contact was defined as a primary care contact on a given calendar date with either a nurse, general physician (GP) or other healthcare professional that were considered as COPD-related, if the most prominent signs and symptoms the participant was presenting were as a direct result of the participant's COPD, as per Readcodes recorded in the patients electronic health record (EHR). The analysis method was General Linear Model assuming an underlying negative binomial distribution with a log-link function and logarithm of time on treatment as an offset variable and adjusted for randomised treatment, baseline COPD maintenance therapy per randomisation stratification, number of moderate/severe COPD exacerbations in the previous year to randomisation and smoking status at baseline.
Time Frame: Up to 54 weeks
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Contacts per participant per year
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Contacts per participant per year | 2.46 [2.34 to 2.58] | 2.42 [2.30 to 2.53]
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p = 0.622, Generalized linear model; Adjusted treatment ratio = 0.98, 95% CI 2-sided [0.92 to 1.05]

7. Secondary Outcome: Number of All Secondary Care Contacts Expressed Using Least Square Mean
Description: A secondary care contact was defined as an inpatient admission or a specialist outpatient visit or an A&E contact. A participant with an A&E contact and subsequent inpatient admission was considered to have had two healthcare contacts. In the situation where inpatient admissions were recorded at two hospitals on the same day, this was counted as a single secondary care contact. The analysis method was General Linear Model assuming an underlying negative binomial distribution with a log-link function and logarithm of time on treatment as an offset variable and adjusted for randomised treatment, baseline COPD maintenance therapy per randomization stratification, number of moderate/severe COPD exacerbations in the previous year to randomization and smoking status at baseline.
Time Frame: Up to 54 weeks
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Contacts per participant per year
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Contacts per participant per year | 9.36 [8.74 to 10.02] | 9.81 [9.17 to 10.51]
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p = 0.336, Generalized Linear Model; Adjusted treatment ratio = 1.05, 95% CI 2-sided [0.95 to 1.15]

8. Secondary Outcome: Number of All Primary Care Contacts Expressed Using Least Square Mean
Description: A primary care contact was defined as contact with a either a nurse, general practitioner, or other healthcare professional. The analysis method was General Linear Model assuming an underlying negative binomial distribution with a log-link function and logarithm of time on treatment as an offset variable and adjusted for randomised treatment, baseline COPD maintenance therapy per randomisation stratification, number of moderate/severe COPD exacerbations in the previous year to randomisation and smoking status at baseline.
Time Frame: Up to 54 weeks
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Contacts per participant per year
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Contacts per participant per year | 18.88 [18.06 to 19.74] | 21.20 [20.27 to 22.16]
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p < 0.001, Generalized Linear Model; Adjusted treatment ratio = 1.12, 95% CI 2-sided [1.05 to 1.20]

9. Secondary Outcome: Time to an Event of Discontinuation of Initial Therapy Occurring in a Year
Description: Initial therapy was defined as the treatment that the subject was randomised to at randomisation. Discontinuation of initial therapy was defined as any modification of initial therapy. These included stepping up, stepping down or switching to another class/class combination, or withdrawal from the study. Switching within the same drug class did not count unless participant switched from FF/VI to a different ICS/LABA. The analysis method was a Cox proportional hazards model adjusted for randomized treatment. The probability of discontinuation of initial therapy was measured from the date of randomisation (i.e., exposure start date) to the date of discontinuation of initial therapy to which the participant was randomized, or date of treatment termination (Visit 6 or early withdrawal visit) for participants who completed the study without discontinuing the initial therapy (censored). Number of participants with event is presented.
Time Frame: Up to 364 days
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 219 | 374
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p < 0.001, Cox proportional hazards model; Hazard Ratio (HR) = 1.89, 95% CI 2-sided [1.60 to 2.23] — A hazard ratio <1 indicates a lower risk with FF/VI compared with Usual Care

10. Secondary Outcome: Time to the Addition of a Further COPD Controller Medication Occurring in a Year
Description: The date of an event for addition of a further COPD controller medication was defined as the exposure start date of the first modified treatment medication that included a new COPD maintenance therapy of a new class of drug (to the initial therapy) during the study treatment period, as collected on the investigational product page of the eCRF. Participants who did not add any COPD controller medication during the study were censored at the end of the treatment period (Day 364). This was equivalent to stepping up, defined as the addition of at least one new class of drug. The probability of an event was measured from the date of randomisation (i.e., treatment initiation) to the date of a change event. The analysis method was a Cox proportional hazards model adjusted for randomized treatment. Number of participants with event is presented.
Time Frame: Up to 364 days
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 142 | 72
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p < 0.001, Cox proprotional hazards model; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.37 to 0.66] — A hazard ratio <1 indicates a lower risk with FF/VI compared with Usual Care

11. Secondary Outcome: Time to First Moderate/Severe Exacerbations Occurring in a Year
Description: The date of an event for moderate / severe COPD exacerbation was defined as the exacerbation onset date. The analysis method was a Cox proportional hazards model adjusted for randomized treatment. The probability of a first moderate / severe exacerbation was measured from the date of randomisation (i.e., treatment initiation) to the onset date of first moderate or severe COPD exacerbation, as recorded on eCRF, or date of treatment termination (Visit 6 or early withdrawal visit) for participants who completed the study without any moderate or severe exacerbations (censored). Participants who completed the study without a moderate or severe COPD exacerbation and analyses of time to first moderate/severe exacerbation were censored at Day 364. Number of participants with event is presented.
Time Frame: Up to 364 days
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 977 | 947
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p = 0.111, Cox porportional hazards model; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.85 to 1.02] — A hazard ratio <1 indicates a lower risk with FF/VI compared with Usual Care

12. Secondary Outcome: Time to First Moderate/Severe Exacerbations on Initial Therapy Occurring in a Year
Description: The date of an event for moderate / severe COPD exacerbation was defined as the exacerbation onset date. The analysis method was a Cox proportional hazards model adjusted for randomized treatment. The probability of first moderate / severe exacerbation on initial therapy was measured from the date of randomisation (i.e., exposure start date) to the onset date of first moderate or severe COPD exacerbation, or to the date of discontinuation of initial therapy (analysis was censored at date of discontinuation of initial therapy) for participants who completed the study without any moderate or severe exacerbations on initial therapy. Number of participants with event is presented.
Time Frame: Up to 364 days
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 943 | 852
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p = 0.081, Cox porportional hazards model; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.84 to 1.01]

13. Secondary Outcome: Time to First Severe Exacerbations Occurring in a Year
Description: The date of an event for severe exacerbation was defined as the exacerbation onset date. Participants who completed the study without a severe exacerbation were censored. The analysis method was a Cox proportional hazards model adjusted for randomized treatment.
  The probability of first severe exacerbation was measured from the date of randomisation (i.e., treatment initiation) to the onset date of first severe exacerbation, as recorded on eCRF, or date of treatment termination (Visit 6 or early withdrawal visit) for participants who completed the study without any severe exacerbations (censored). At Day 364, all participants who have not experienced a severe exacerbation are considered censored, regardless of whether their on-treatment phase continues beyond day 364, including those who withdrew early. Number of participants with event is presented.
Time Frame: Up to 364 days
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 97 | 122
Statistical Analysis 1: Comparison: Usual Care vs FF/VI 100 mcg/25 mcg; Test type: Superiority or Other; p = 0.075, Cox proportional hazards model; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.98 to 1.66]

14. Secondary Outcome: Number of Participants With Fatal Serious Adverse Events of Pneumonia
Description: All SAEs included in the AE subgroup of special interest of "pneumonia" were considered as an SAE of pneumonias. A fatal SAE was defined as a SAE with outcome of fatal for study participant. The number of participants with fatal SAEs of pneumonia was assessed over 14 months.
Time Frame: Upto 58 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 13 | 13

15. Secondary Outcome: Number of Participants With Non-serious Adverse Drug Reactions (ADR)
Description: The number of participants with non-serious ADRs was assessed for up to 54 weeks. An ADR is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, for which there is a reasonable possibility that the untoward occurrence is causally related to the medicinal product. A non-serious ADR included one of the following: exacerbation of chronic or intermittent pre-existing condition; signs, symptoms, or the clinical sequelae of a suspected interaction; signs, symptoms, or new conditions detected or diagnosed after study treatment administration.
Time Frame: Up to 54 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 88 | 192

16. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: SAEs assessed included medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a significant medical event in the investigator's judgment, or is an event of possible drug-induced liver injury with hyperbilirubinaemia. SAEs were includes if the onset date was on or after the treatment start date and on or before the treatment stop date. However, the window for an SAE of pneumonia was longer and included 28 days post study treatment stop date.
Time Frame: Up to 56 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 383 | 404

17. Secondary Outcome: Number of Participants With Serious Adverse Drug Reactions
Description: A serious adverse drug reactions (SADR) is any untoward medical occurrence suspected to be medicinal product-related that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Upto 12 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Number analyzed (Participants) | 1403 | 1396
Participants | 10 | 23

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs; from Visit 1) and non-serious adverse drug reactions (from Visit 2) were collected from study medication start until the end of treatment (up to Visit 6 or withdrawal, ie, approximately 54 weeks)
Arm/Group | Usual Care | FF/VI 100 mcg/25 mcg
Serious Adverse Events (participants affected / at risk) | 383/1403 | 404/1396
Other Adverse Events (participants affected / at risk) | 40/1403 | 56/1396
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=1403) | FF/VI 100 mcg/25 mcg (N=1396)
Pneumonia (Infections and infestations) | 81 | 89
Infective exacerbation of chronic obstructive airway disease (Infections and infestations) | 47 | 50
Cellulitis (Infections and infestations) | 9 | 14
Lower respiratory tract infection (Infections and infestations) | 10 | 12
Urinary tract infection (Infections and infestations) | 12 | 9
Sepsis (Infections and infestations) | 10 | 9
Gastroenteritis (Infections and infestations) | 4 | 3
Urosepsis (Infections and infestations) | 1 | 4
Abdominal sepsis (Infections and infestations) | 2 | 2
Biliary sepsis (Infections and infestations) | 2 | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 3
Gastroenteritis viral (Infections and infestations) | 2 | 2
Osteomyelitis (Infections and infestations) | 3 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 1
Anal abscess (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 2
Endocarditis (Infections and infestations) | 2 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 2
Ophthalmic herpes zoster (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Abscess limb (Infections and infestations) | 0 | 1
Abscess oral (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Herpes zoster meningoencephalitis (Infections and infestations) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 1
Mycetoma mycotic (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Septic embolus (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Viral labyrinthitis (Infections and infestations) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 70 | 86
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 24 | 15
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 29 | 27
Acute myocardial infarction (Cardiac disorders) | 9 | 13
Cardiac failure (Cardiac disorders) | 11 | 10
Acute coronary syndrome (Cardiac disorders) | 12 | 5
Angina pectoris (Cardiac disorders) | 9 | 5
Cardiac failure congestive (Cardiac disorders) | 5 | 6
Angina unstable (Cardiac disorders) | 4 | 5
Myocardial infarction (Cardiac disorders) | 3 | 6
Myocardial ischaemia (Cardiac disorders) | 3 | 4
Left ventricular dysfunction (Cardiac disorders) | 4 | 2
Atrial flutter (Cardiac disorders) | 2 | 3
Cor pulmonale (Cardiac disorders) | 2 | 3
Ventricular tachycardia (Cardiac disorders) | 3 | 2
Left ventricular failure (Cardiac disorders) | 3 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 4
Arrhythmia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 2 | 1
Right ventricular failure (Cardiac disorders) | 0 | 3
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 2
Cardiogenic shock (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Trifascicular block (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 15
Rib fracture (Injury, poisoning and procedural complications) | 9 | 5
Radius fracture (Injury, poisoning and procedural complications) | 5 | 8
Head injury (Injury, poisoning and procedural complications) | 2 | 8
Hand fracture (Injury, poisoning and procedural complications) | 4 | 4
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 5
Ankle fracture (Injury, poisoning and procedural complications) | 5 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 4
Alcohol poisoning (Injury, poisoning and procedural complications) | 4 | 2
Foot fracture (Injury, poisoning and procedural complications) | 2 | 4
Intentional overdose (Injury, poisoning and procedural complications) | 2 | 4
Overdose (Injury, poisoning and procedural complications) | 3 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 3 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 3
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 | 0
Cardiac valve rupture (Injury, poisoning and procedural complications) | 0 | 1
Chemical injury (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Open fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 0 | 1
Syncope (Nervous system disorders) | 10 | 11
Transient ischaemic attack (Nervous system disorders) | 9 | 5
Ischaemic stroke (Nervous system disorders) | 6 | 3
Seizure (Nervous system disorders) | 4 | 3
Cerebrovascular accident (Nervous system disorders) | 5 | 1
Cerebrovascular disorder (Nervous system disorders) | 2 | 2
Cerebral infarction (Nervous system disorders) | 1 | 2
Brain injury (Nervous system disorders) | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 1
VIth nerve paralysis (Nervous system disorders) | 0 | 2
Vocal cord paresis (Nervous system disorders) | 0 | 2
Basal ganglia infarction (Nervous system disorders) | 1 | 0
Brain mass (Nervous system disorders) | 1 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0
Carotid sinus syndrome (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Dementia with Lewy bodies (Nervous system disorders) | 0 | 1
Drug withdrawal convulsions (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Meningism (Nervous system disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Radiculitis brachial (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 10
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid body tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 16 | 23
Renal impairment (Renal and urinary disorders) | 7 | 10
Urinary retention (Renal and urinary disorders) | 7 | 8
Chronic kidney disease (Renal and urinary disorders) | 5 | 2
Haematuria (Renal and urinary disorders) | 3 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 2 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 1
Sterile pyuria (Renal and urinary disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Haematemesis (Gastrointestinal disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Gastritis (Gastrointestinal disorders) | 2 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 4
Colitis ischaemic (Gastrointestinal disorders) | 1 | 3
Colitis (Gastrointestinal disorders) | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Diverticulum (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Coeliac disease (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyskinesia oesophageal (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric dysplasia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatic insufficiency (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 7
Electrolyte imbalance (Metabolism and nutrition disorders) | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 6
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 5
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4
Gout (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Liver function test abnormal (Investigations) | 6 | 15
Renal function test abnormal (Investigations) | 9 | 12
Electrocardiogram QT prolonged (Investigations) | 2 | 2
International normalised ratio increased (Investigations) | 2 | 1
Weight decreased (Investigations) | 1 | 2
Haemoglobin decreased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood electrolytes abnormal (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 9
Aortic aneurysm (Vascular disorders) | 3 | 3
Aortic stenosis (Vascular disorders) | 2 | 4
Haematoma (Vascular disorders) | 3 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 4
Hypotension (Vascular disorders) | 3 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 1
Angiodysplasia (Vascular disorders) | 1 | 1
Lymphoedema (Vascular disorders) | 1 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 3
Cholangitis (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 3
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Delirium (Psychiatric disorders) | 2 | 4
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 3
Confusional state (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 3 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 2 | 0
Delirium tremens (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Self-injurious ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 6 | 5
Microcytic anaemia (Blood and lymphatic system disorders) | 4 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1
Chest pain (General disorders) | 8 | 1
Non-cardiac chest pain (General disorders) | 1 | 4
Cyst (General disorders) | 1 | 0
Hypothermia (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Stent-graft endoleak (General disorders) | 0 | 1
Unintentional medical device removal (General disorders) | 1 | 0
Vascular stent occlusion (General disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 2
Blindness unilateral (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 2
Anaphylactic reaction (Immune system disorders) | 0 | 2
Drug hypersensitivity (Immune system disorders) | 2 | 0
Allergic granulomatous angiitis (Immune system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 1
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 2 | 0
Carotid endarterectomy (Surgical and medical procedures) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=1403) | FF/VI 100 mcg/25 mcg (N=1396)
Oral candidiasis (Infections and infestations) | 40 | 56 — In this study, only information regarding non- serious adverse drug reactions (ADRs) and serious adverse events (SAEs) were detected, documented and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.